CLINICAL TRIAL: NCT02331459
Title: Effect of a Multicomponent Training Intervention on Cognition, Mood, and Function in a Controlled Population of Community-dwelling Frail Elderly Patients.
Brief Title: Training Intervention in a Controlled Population of Frail Elderly
Acronym: EMTIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de la Ribera (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Francisco Jose Tarazona-Santabalbina, MD PhD, Hospital de la Ribera
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HULR-EMTIFE-2013-1
Record Dates: First submitted 2015-01-03; First posted 2015-01-06 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Physical Activity
Keywords: mood; cognitive state; physical activity; frailty
MeSH Terms: conditions — Motor Activity; Frailty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Multicomponent training intervention :
  3 sessions a week of 45 minutes of resistance activity (24 weeks) 2 sessions a week of 45 minutes of strength training (24 weeks) 5 sessions a week of 15 minutes of proprioceptive training (24 weeks)
  Interventions: Other: Multicomponent training intervention; Other: Nutritional intervention
- Control group (Placebo Comparator): Normal routine during 24 weeks.
  Interventions: Other: Nutritional intervention

INTERVENTIONS:
Other: Multicomponent training intervention — Intervention characteristics: 24weeks, 5days/week, 60min/session Day 1, 3 and 5 15 min (a) 40 min (b) 5 min (d) Day 2 and 4 15 min (a) 40 min (c) 5 min (d)
  Legend:
  min. =minutes a = Proprioception exercises, postural sway and dynamic balance, coordination and flexibility of the lumbo-pelvic area b = Aerobic training 65% maximal Heart rate c = Strength training arms and legs d = Stretching
  Arms: Intervention group
Other: Nutritional intervention — Enrolled patients will receive nutritional information on optimal daily energy intake, ensuring at least a daily protein intake of 1 g. of by kg of weight.
  Calcium plus vitamin D (total amount 1200 mg calcium plus 800 IU of vitamin D) Vitamin D will be provided if calcidiol (Cldl) blood levels are lower than 30 ng/ml.
  Cldl 20-29 ng/dl it will provide calciferol 20.000 IU every 15 days (3 months) Cldl 10-19 ng/dl it will provide calciferol 20.000 IU every 10 days (3 months) Cldl 1-9 ng/dl it will provide calciferol 20.000 IU every 7 days (3 months)

SUMMARY:
Exercise has a beneficial role in geriatric patients categorized as frail. Nevertheless, it is not known physical training pattern more beneficial for these patients. The reasons for heterogeneity and lack of consistency of the results described by published intervention programs may be the diversity of isolated - resistance, endurance or proprioceptive trainings - or a combination of them. There are no studies with a combined program of this three kinds of physical training.

The objective of this study is to know if a multicomponent physical training program during 180 days in dwelling-community frail geriatric patients can improve scores on functional, activities of daily living, mood, cognitive and quality of life scales and producing changes in blood levels of biological and genetic markers.

DETAILED DESCRIPTION:
At the start of recruitment, a comprehensive geriatric assessment will be developed in enrolled patients of both groups. After this assessment and before starting the physical training in intervention group, a nutritional intervention will be provided in patients of both groups :

Enrolled patients will receive nutritional information on optimal daily energy intake, ensuring at least a daily protein intake of 1 g. of by kg of weight.

As well as, calcium and vitamin D will be provided if calcidiol blood levels are lower than 30 ng/ml.

Calcidiol blood value between 20-29 ng/dl it will provide calcium + vitamin D (total amount 1200 mg calcium plus 800 IU of vitamin D) daily and calciferol 20.000 IU every 15 days (3 months)

Calcidiol blood value between 10-19 ng/dl it will provide calcium + vitamin D (total amount 1200 mg calcium plus 800 IU of vitamin D) daily and calciferol 20.000 IU every 10 days (3 months)

Calcidiol blood value between 1-9 ng/dl it will provide calcium + vitamin D (total amount 1200 mg calcium plus 800 IU of vitamin D) daily and calciferol 20.000 IU every 7 days (3 months)

After nutritional intervention, intervention group will start a multicomponent training intervention during 180 days Intervention characteristics: 24weeks, 5days/week, 60min/session Day 1, 3 and 5 15 min (a) 40 min (b) 5 min (d) Day 2 and 4 15 min (a) 40 min (c) 5 min (d)

Legend:

min. =minutes a = Proprioception exercises, postural sway and dynamic balance, coordination and flexibility of the lumbo-pelvic area b = Aerobic training 65% HRmax c = Strength training arms and legs d = Stretching Characteristics of the strength training Month 1 Week 1 25% 1-RM 1x30 r Week 2 25% 1-RM 2x30 r Week 3-4 25% 1-RM 3x30 r Month 2 Week 1-4 25% 1-RM 3x30 r Month 3 Week 1 50% 1-RM 1x15 r Week 2 50% 1-RM 2x10 r Week 3-4 50% 1-RM 3x8 r Month 4 Week 1-4 50% 1-RM 3x8 r Month 5 Week 1 75% 1-RM 1x15 r Week 2 75% 1-RM 2x10 r Week 3-4 75% 1-RM 3x8 r Month 6 Week 1-4 75% 1-RM 3x8 r

Legend:

1-RM: One-repetition maximum r: repetitions

Monthly, enrolled frail elderly patients will be evaluated. 6 minutes walking test, timed up and go test, bilateral hand grip, Barthel index, Tinetti balance assessment tool, Mini-mental state examination, short-MNA (Mini Nutritional Assessment ), lean and fat mass measures with impedanciometer and number of visits to general practitioner, emergency room and hospital admission were recorded.

After follow up period a new comprehensive geriatric assessment will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. - Dwelling-community subjects
2. - Age 70 years old and older
3. Frail geriatric patient according to the Cardiovascular Health Study (CHS) Frailty Phenotype
4. Gait speed less than 0.8 m/s.

Exclusion Criteria:

1. - Life expectancy less than 6 months for any clinical reason (we considered criteria of a life expectancy less than 6 months 7 c-7 d global deterioration degree on GDS (Global Deterioration Scale)-FAST (Functional Assessment Staging ) scale in patients with dementia; severe disabilities considered as score less than 15 points in Barthel index and left ventricular ejection fraction equal or less than 20%)
2. - Hospital Admission in the last 3 months for any clinical reason
3. - oncologic patients in chemotherapy or radiotherapy active treatment
4. - Major surgery in the last 6 months
5. - First-degree centenary relatives in the two previous generations
6. - Ischemic coronary event in the last 12 months
7. Institutionalized subjects
8. Impossibility of displacement to the Health Center by themselves.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Activities of daily living. | Day 0 and Day 180 (plus or minus 3 days)
  The primary study endpoint is the change from baseline to the end of the intervention, and the change between the intervention group and the control group, in score of Barthel Activities of Daily Living Index and the Lawton Instrumental Activities of Daily Living Scale

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | Day 0 and Day 180 (plus or minus 3 days)
  Change from baseline to the end of the intervention, and the change between the intervention group and the control group.
Short Physical Performance Battery and Physical Performance Test | Day 0 and Day 180 (plus or minus 3 days)
  Change from baseline to the end of the intervention, and the change between the intervention group and the control group.

OTHER OUTCOMES:
Geriatric Depression Scale | Day 0 and Day 180 (plus or minus 3 days)
  Change from baseline to the end of the intervention, and the change between the intervention group and the control group.
Quality of life: EuroQol-5D | Day 0 and Day 180 (plus or minus 3 days)
  Change from baseline to the end of the intervention, and the change between the intervention group and the control group.
Composite effect of a multicomponent training intervention on systemic biomarkers of frailty | Day 0 and Day 180 (plus or minus 3 days)
  * Plasma malondialdehyde (High performance liquid chromatography)
  * Plasma oxidized proteins (Western blotting)
  * serum interleukin (IL)-6 and tumor necrosis factor (TNF)-α (ELISA Kits)
  * Plasma GDF-11 (Western Blotting)
  * Plasma Meterorin-like (ELISA kit)

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Pérez-Ros, PhD, Study Chair — Catholic University of Valencia San Vicente Mártir; Francisco Martínez-Arnau, PhD, Study Chair — University of Valencia; Jose Vina, MD,PhD, Study Director — Univeristy of Valencia; Carmen Gómez-Cabrera, PhD, Study Chair — University of Valencia; Francisco J Tarazona-Santabalbina, MD, PhD, Principal Investigator — Hospital de la Ribera
Locations (1):
- Hospital Universitario de la Ribera, Alzira, Valéncia, Spain

REFERENCES:
- [Derived] Tarazona-Santabalbina FJ, Gomez-Cabrera MC, Perez-Ros P, Martinez-Arnau FM, Cabo H, Tsaparas K, Salvador-Pascual A, Rodriguez-Manas L, Vina J. A Multicomponent Exercise Intervention that Reverses Frailty and Improves Cognition, Emotion, and Social Networking in the Community-Dwelling Frail Elderly: A Randomized Clinical Trial. J Am Med Dir Assoc. 2016 May 1;17(5):426-33. doi: 10.1016/j.jamda.2016.01.019. Epub 2016 Mar 3. PMID 26947059